CLINICAL TRIAL: NCT02677870
Title: The Effectiveness of High-Dose Synthetic BH4 (Saproterin Dihydrochloride or "Kuvan") in Amish PKU Patients
Brief Title: The Effectiveness of Kuvan in Amish PKU Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UHCMC IRB#
Record Dates: First submitted 2016-01-26; First posted 2016-02-09 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Phenylketonuria
Keywords: Saproterin dihydrochloride; Kuvan; Amish
MeSH Terms: conditions — Phenylketonurias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Diet treatment (Other): In part 1 of the study, patients will not receive any medication. Each patient will DIET treatment alone. They will maintain a stable, Phe restricted diet (including formula) that is consistent with their diet at the time of enrollment. This will be monitored by food diaries kept for 3 days of each week. Based on these diaries, average weekly Phe intake and Phe tolerance will be calculated and recorded.
  Interventions: Other: Diet treatment
- Standard dose saproterin dihydrochloride (Active Comparator): Study numbers will be randomized into "standard-dose saproterin dihydrochloride (Kuvan)" or "high-dose saproterin dihydrochloride (Kuvan) " groups (treatment group A or treatment group B). Both groups will receive a trial of both standard and high dose saproterin dihydrochloride before the end of the study. Standard-dose saproterin dihydrochloride will be 20mg/kg (rounded up to the nearest 100mg) provided in the form of 100mg tablets. Dosing of the tablets will be unidentifiable to patients. Medication will be given orally once daily.
  Interventions: Drug: saproterin dihydrochloride; Other: Diet treatment
- High dose saproterin dihydrochloride (Experimental): Study numbers will be randomized into "standard-dose saproterin" or "high-dose saproterin" groups (treatment group A or treatment group B). Both groups will receive a trial of both standard and high dose saproterin dihydrochloride before the end of the study. Goal high-dose saproterin dihydrochloride dosing will be 40mg/kg (rounded up to the nearest 500mg), provided in the form of pre-packaged 500mg packets of powder. Labeled dosing on these packets will be covered by the investigational drug pharmacy and unidentifiable to patients. Dosing of the tablets will be unidentifiable to patients. Medication will be given orally once daily.
  Interventions: Drug: saproterin dihydrochloride; Other: Diet treatment

INTERVENTIONS:
Drug: saproterin dihydrochloride — The drug will be given as described in the arm/group descriptions.
  Other Names: Kuvan treatment
  Arms: High dose saproterin dihydrochloride; Standard dose saproterin dihydrochloride
Other: Diet treatment — Patients will maintain a stable, Phe restricted diet (including formula) that is consistent with their diet at the time of enrollment. This will be monitored by food diaries kept for 3 days of each week.

SUMMARY:
The purpose of this study is to determine if Amish patients with PKU show responsiveness after a high dose, prolonged Saproterin trial. The population of interest has a high frequency of a specific splice site mutation, the 1066-11G>A mutation. This splice site mutation activates a cryptic splice site resulting in an in frame insertion of 9 nucleotides preceding exon 11. This leads to protein conformational changes and abrogation of function. Previous studies of this genotype have indicated <1% residual activity of the PAH enzyme and an insignificant responsiveness to Saproterin. However, in this specific study Phe levels were evaluated only over 24 hours after a single-dose BH4 challenge at the standard dose of 20mg/kg.

Based on new clinical information, the investigators hypothesize that if given a prolonged trial of Saproterin at a higher dose, Amish patients with PKU, specifically those homozygous for the c.1066-11G>A mutation, will have a significant reduction in Phe levels or an increase in Phe tolerance and/or improvement in executive functioning and quality of life.

DETAILED DESCRIPTION:
Phenylketonuria (PKU) is caused by a deficiency of the enzyme phenylalanine hydroxylase (PAH). PAH is responsible for the rate limiting step in phenylalanine catabolism. This reaction is dependent on tetrahydrobiopterin (BH4). BH4 is a catalytic cofactor for the enzyme PAH. Supplementation with synthetic BH4 (saproterin dihydrochloride or KuvanTm) has been shown to activate residual PAH activity and lower Phe levels in certain patients. It may also have a chaperone effect by binding abnormal PAH protein and decreasing its degradation. Saproterin is an approved oral drug developed to reduce blood Phenylalanine (Phe) levels and increase Phe tolerance in BH4 responsive patients with hyperphenylalaninemia.

Certain genotypes have been found to be good predictors of Saproterin responsiveness; however, these correlations are imperfect. Therefore the standard of care is to perform a trial of Saproterin therapy to assess responsiveness in every PAH patient regardless of genotype. Currently this recommendation does not include patients with two null mutations.

The purpose of this study is to determine if Amish patients with PKU show responsiveness after a high dose, prolonged Saproterin trial. The population of interest has a high frequency of a specific splice site mutation, the 1066-11G>A mutation. This splice site mutation leads to protein conformational changes and abrogation of function. Previous studies of this genotype have indicated <1% residual activity of the PAH enzyme and an insignificant responsiveness to Saproterin. However, in this specific study Phe levels were evaluated only over 24 hours after a single-dose BH4 challenge at the standard dose of 20mg/kg.

Recently, observation in several Amish patients suggests some promise that these patients may be responsive to Saproterin after a longer trial of the medication (Personal comment - Samuel Yang, MD). In addition, studies evaluating PAH enzyme activity in these patients, have found evidence that this genotype may need higher cofactor concentrations for optimal enzyme activity and therefore may require a higher dose of Saproterin then the currently recommended 20mg/kg (9). To date, no formal clinical trial has been done.

To answer the question of whether this genotype is responsive to Saproterin at higher doses, over a prolonged period, the investigators propose a randomized clinical trial comparing blood Phe levels in patients treated with standard-dose Saproterin to those treated with high-dose Saproterin. The results of this study could reveal a new population of Saproterin responsive PKU patients. This could call into question other null mutations of the PAH gene and their responsiveness to Saproterin. This may lead to the investigation of genotypes previously thought to be unresponsive to Saproterin. Further, diet treatment alone has proven to be difficult for the Amish population for cultural and economic reasons.

This study will include patients from three local centers with the potential of a fourth, out of state, center participating. All patients will be enrolled through University Hospitals Case Medical Center. Consent will be obtained over the phone or in person.

* Amish patients from University Hospitals Case Western Reserve/Rainbow Babies and Children's Hospital/Center for Human Genetics
* Amish patients from Akron Children's hospital in Akron, Ohio
* Amish patients from The Center for Children with Special Needs (DDC clinic), Middlefield, Ohio
* Patients from Shodair Children's Hospital in Helena, Montana. These patients may be recruited if more patients are required to meet our enrollment goal.

Study patients will present to their preferred clinic for 5 office visits. Initial testing/Part 1: length 4 weeks

Recruited patients will present to clinic for part 1 of the study. After informed consent is obtained, molecular genetic testing will be performed. Testing will include sequence analysis of the PAH gene. This testing is necessary to identify the specific genotypes present in each patient. The investigators expect the majority of this population to be homozygous or heterozygous for the above described splice site mutation. Any patients found to have one (or no) identifiable mutations after sequencing will not be included in the study. Genotypes will be grouped and analyzed separately at the conclusion of the study. Patients who do not wish to undergo genetic testing will not be included in the study.

Each patient will also have an initial blood Phe level drawn in the form of a dried blood spot on filter paper card that will be supplied by the testing company. All Phe testing will be performed in a Clinical Laboratory Improvement Amendment (CLIA) certified laboratory at The Clinic for Special Children in Strasburg, PA.

Baseline assessment tools (BRIEF, PKU-QOL) will also be performed at this initial visit. Patients will be given a unique study number by our investigational drug pharmacy and will begin part 1 of the study as described below.

In part 1 of the study, patients will not receive any medication. Each patient will be treated with diet alone. Patients will maintain a stable, Phe restricted diet (including formula) that is consistent with their diet at the time of enrollment. This will be monitored by food diaries kept for 3 days of each week. Specifically, patients will be expected to keep diaries for the 3 consecutive days leading up to blood draw. Based on these diaries, average weekly Phe intake and Phe tolerance will be calculated and recorded. Patients will also complete a food frequency tool, which will be reviewed at part 1, 2 and 3's initial visit. We will use all of the tools above, plus allow patients regular access to our dietician in order to encourage the maintenance of a stable diet.

Blood Phe concentration will be measured weekly (each Monday) by blood spot cards. Patients will not require weekly clinic visits to have Phe levels drawn. Blood spot cards will be performed at their home and then mailed to the reference laboratory. In order to teach and enable patients to become comfortable performing their own blood spots at home, nursing staff (from the DDC clinic) will travel to each patient's house weekly for part 1 of the study (total of 3 home blood spots). For parts 2 and 3 of the study, those patients and families who are able, will perform their own blood spots at home. Those families who remain uncomfortable performing their own blood spots will continue to have their blood spots collected by home nursing.

Initial visit:

* Venous blood draw for PAH gene sequencing
* Baseline Phe level by dried blood spot card in office
* Executive functioning and quality of life assessment tools (BRIEF, PKU-QOL) given
* Baseline diet information collected and recorded. Average weekly Phe calculated, Phe tolerance calculated.
* Food frequency tool completed and reviewed.

Blood Phe values and Phe tolerance from part 1 of the study (on diet treatment alone) will be compared to blood Phe values and Phe tolerance from parts 2 and 3, on low-dose and high-dose treatment.

Part 2: length - 4 weeks

Study numbers will be randomized into "standard-dose Saproterin" or "high-dose Saproterin" groups (treatment group A or treatment group B). The investigational drug pharmacy will provide study patients with their medication in kits, at the beginning of each treatment period. Goal high-dose Saproterin dosing will be 40mg/kg (rounded up to the nearest 500mg), provided in the form of pre-packaged 500mg packets of powder. Labeled dosing on these packets will be covered by the investigational drug pharmacy and unidentifiable to patients. Standard-dose Saproterin will be 20mg/kg (rounded to the nearest 100mg) provided in the form of 100mg tablets. Dosing of the tablets will be unidentifiable to patients. Medication will be given orally once daily.

Initial part 2 visit: after 4 week diet only period

* Food diaries collected for the previous 4 weeks (3 per week). Average weekly Phe calculated, Phe tolerance calculated.
* Food frequency tool completed and reviewed.
* Baseline Phe level drawn by dried blood spot card in office
* Executive functioning and quality of life assessment tools (BRIEF, PKU-QOL) given
* Provided with medication kits (high or standard-dose, 4 week supply)

Final part 2 visit: after 4 weeks of treatment

* Food diaries collected for the previous 4 weeks (3 per week). Average weekly Phe calculated, Phe tolerance calculated.
* Executive functioning and quality of life assessment tools (BRIEF, PKU-QOL) given
* Empty medication bottles/packet kits collected from each patient to assess compliance
* Review of any potential adverse events

This is the end of part 2. There will then be a 2 week "wash out period" where patients receive no treatment. The length of this washout period was determined based on the mean elimination half-life of saproterin and previous clinical trials. The mean elimination half-life of saproterin ranges from 3.9 to 17 hours. In previous trials, washout periods have consisted of 7 and 30 days. No efficacy assessments have been performed to differentiate or support one washout period over the other (BioMarin Pharmaceuticals, Inc. Data on file). Based on the elimination range above, we determined that a two week washout period is sufficient. Patients should maintain their steady diet during this time.

Part 3: length - 4 weeks The cross-over will occur between treatment groups: A to B and B to A.

Initial part 3 visit: after 2 week washout period

* Food diaries collected for the previous 2 weeks (3 per week). Average weekly Phe calculated, Phe tolerance calculated.
* Food frequency tool completed and reviewed.
* Baseline Phe level performed by dried blood spot card in office
* Executive functioning and quality of life assessment tools (BRIEF, PKU-QOL) given
* Provided with medication kits (high or standard-dose, 4 week supply)
* Review of any potential adverse events

Final part 3 visit: after 4 weeks of treatment

* Food diaries collected for the previous 4 weeks (3 per week)
* Executive functioning and quality of life assessment tools (BRIEF, PKU-QOL) given
* Empty medication bottles/ kits collected from each patient to assess compliance
* Review of any potential adverse events

During all parts, patients will maintain a stable, Phe restricted diet including formula (same diet as in part 1 of the study). All Phe levels will be blinded and researchers will not have access to them until the conclusion of the study. At the conclusion of the study, after all data have been analyzed, a complete list of blood Phe levels obtained during the study (both on high and low-dose treatment) will be sent to each patient's primary metabolic physician. Physicians can then discuss long term Saproterin treatment with their patients based on their Phe levels.

The study will conclude after all parts are complete and groups A and B have both received a trial of high and standard-dose Saproterin. All medication will be discontinued at this time.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of PKU with the following:
* Age of at least 2 years or older
* Baseline Phe level of > 360 umol/L
* Willing to maintain a stable diet
* Patient or guardian are willing and able to provide written, signed informed consent after the nature of the study has been explained and prior to any research-related procedures
* Are willing to comply with all study procedures
* Two identifiable mutations found on PAH gene sequencing
* Any patients already taking Saproterin (or have taken in the past), must have a treatment end date at least 14 days prior to Day 1 of the study.

Exclusion Criteria:

* Any patient currently taking Saproterin who has taken the medication at any point in the 14 days prior to Day 1 of the study
* Under 2 years of age
* Unwilling to maintain a stable diet
* Patients with baseline Phe levels < 360 umol/L
* Patients unable to comply with all study procedures
* Patients unable to provide written, signed informed consent
* One (or no) identifiable mutations found on PAH gene sequencing

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-22 (Actual); Primary Completion 2018-11-20 (Actual); Study Completion 2019-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori-Anne P Schillaci, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wang H, Nye L, Puffenberger E, Morton H. Phenylalanine hydroxylase deficiency exhibits mutation heterogeneity in two large old order Amish settlements. Am J Med Genet A. 2007 Aug 15;143A(16):1938-40. doi: 10.1002/ajmg.a.31852. No abstract available. PMID 17630668
- [Background] Dobrowolski SF, Heintz C, Miller T, Ellingson C, Ellingson C, Ozer I, Gokcay G, Baykal T, Thony B, Demirkol M, Blau N. Molecular genetics and impact of residual in vitro phenylalanine hydroxylase activity on tetrahydrobiopterin responsiveness in Turkish PKU population. Mol Genet Metab. 2011 Feb;102(2):116-21. doi: 10.1016/j.ymgme.2010.11.158. Epub 2010 Nov 18. PMID 21147011
- [Background] Dworniczak B, Aulehla-Scholz C, Kalaydjieva L, Bartholome K, Grudda K, Horst J. Aberrant splicing of phenylalanine hydroxylase mRNA: the major cause for phenylketonuria in parts of southern Europe. Genomics. 1991 Oct;11(2):242-6. doi: 10.1016/0888-7543(91)90129-3. PMID 1769645
- [Background] Karacic I, Meili D, Sarnavka V, Heintz C, Thony B, Ramadza DP, Fumic K, Mardesic D, Baric I, Blau N. Genotype-predicted tetrahydrobiopterin (BH4)-responsiveness and molecular genetics in Croatian patients with phenylalanine hydroxylase (PAH) deficiency. Mol Genet Metab. 2009 Jul;97(3):165-71. doi: 10.1016/j.ymgme.2009.03.009. Epub 2009 Apr 1. PMID 19394257
- [Background] Zurfluh MR, Zschocke J, Lindner M, Feillet F, Chery C, Burlina A, Stevens RC, Thony B, Blau N. Molecular genetics of tetrahydrobiopterin-responsive phenylalanine hydroxylase deficiency. Hum Mutat. 2008 Jan;29(1):167-75. doi: 10.1002/humu.20637. PMID 17935162
- [Background] Keil S, Anjema K, van Spronsen FJ, Lambruschini N, Burlina A, Belanger-Quintana A, Couce ML, Feillet F, Cerone R, Lotz-Havla AS, Muntau AC, Bosch AM, Meli CA, Billette de Villemeur T, Kern I, Riva E, Giovannini M, Damaj L, Leuzzi V, Blau N. Long-term follow-up and outcome of phenylketonuria patients on sapropterin: a retrospective study. Pediatrics. 2013 Jun;131(6):e1881-8. doi: 10.1542/peds.2012-3291. Epub 2013 May 20. PMID 23690520
- [Background] Waisbren S, White DA. Screening for cognitive and social-emotional problems in individuals with PKU: tools for use in the metabolic clinic. Mol Genet Metab. 2010;99 Suppl 1:S96-9. doi: 10.1016/j.ymgme.2009.10.006. PMID 20123479
- [Background] Regnault A, Burlina A, Cunningham A, Bettiol E, Moreau-Stucker F, Benmedjahed K, Bosch AM. Development and psychometric validation of measures to assess the impact of phenylketonuria and its dietary treatment on patients' and parents' quality of life: the phenylketonuria - quality of life (PKU-QOL) questionnaires. Orphanet J Rare Dis. 2015 May 10;10:59. doi: 10.1186/s13023-015-0261-6. PMID 25958326
- See also: PKU database with known mutations and their responsiveness after Kuvan trial. Length of trial performed is also listed on website. — http://www.biopku.org/biopku

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 7/7 of the patients that were recruited were randomized and completed the study.
Groups:
- Diet tx, Standard Dose Saproterin, Wash, High Dose Saproterin: Enrolled patients with PKU received diet treatment only for 4 weeks. During this portion, no medication was administered and they followed their baseline low protein diet.
  They were then were randomized into standard dose Saproterin dihydrochloride(20 mg/kg/day). They completed 4 weeks of treatment with dosing above being administered once per day.
  There was then a 2 week washout period with no intervention.
  They were then treated with high dose Saproterin dihydrochloride (40 mg/kg/day). They completed 4 weeks of treatment with dosing above being administered once per day.
- Diet, High Dose Saproterin, Wash, Standard Dose Saproterin: Enrolled patients with PKU received diet treatment only for 4 weeks. During this portion, no medication was administered and they followed their baseline low protein diet.
  They were then were randomized into high dose Saproterin dihydrochloride (40 mg/kg/day). They completed 4 weeks of treatment with dosing above being administered once per day.
  There was then a 2 week washout period with no intervention.
  They were then treated with standard dose Saproterin dihydrochloride(20 mg/kg/day). They completed 4 weeks of treatment with dosing above being administered once per day.
Period: Diet Treatment (4 Weeks)
Arm/Group | Diet tx, Standard Dose Saproterin, Wash, High Dose Saproterin | Diet, High Dose Saproterin, Wash, Standard Dose Saproterin
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0
Period: First Saproterin Dihydrochloride tx
Arm/Group | Diet tx, Standard Dose Saproterin, Wash, High Dose Saproterin | Diet, High Dose Saproterin, Wash, Standard Dose Saproterin
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Diet tx, Standard Dose Saproterin, Wash, High Dose Saproterin | Diet, High Dose Saproterin, Wash, Standard Dose Saproterin
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0
Period: Second Saproterin Dihydrochloride tx
Arm/Group | Diet tx, Standard Dose Saproterin, Wash, High Dose Saproterin | Diet, High Dose Saproterin, Wash, Standard Dose Saproterin
Started | 4 | 3
Completed | 4 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients participated in each arm of the trial by the end of this crossover study.
Groups:
- Overall Study: Enrolled patients with PKU received diet treatment only for 4 weeks. Then were randomized into high dose saproterin dihydrochloride (40 mg/kg/day) or low dose saproterin dihydrochloride(20 mg/kg/day).
  They completed 4 weeks of treatment at either dose and then underwent a 2 week washout period without any medication.
  After the washout period, they were crossed over to receive the opposite dose for 4 weeks.
Arm/Group | Overall Study
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 21 [8 to 42]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
Phenylalanine level > 360 umol/L [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With 20% Decrease in Phenylalanine Levels From Baseline (Positive Response)
Description: Subjects will be assessed for plasma Phe concentration by dried blood spot cards during their initial visit (day 1) and every week thereafter. Except during the two week wash-out period where no plasma Phe will be collected. A decrease of plasma Phe levels from baseline by 20% will be considered a positive response.
Time Frame: Baseline, weekly for 4 weeks during diet arm, weekly for 4 weeks during both high and standard dose arms
Population: All participants who completed all 4 weeks in each intervention were included in analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Diet Treatment: Enrolled patients with PKU received diet treatment only for 4 weeks. During this portion, no medication was administered and they followed their baseline low protein diet.
- Standard Dose Saproterin Dihydrochloride: Participants who received Saproterin dihydrochloride at a dose of 20 mg/kg once daily (for 4 weeks) in either the first intervention or second intervention of the study.
- High Dose Saproterin Dihydrochloride: Participants who received Saproterin dihydrochloride at a dose of 40 mg/kg once daily (for 4 weeks) in either the first intervention or second intervention of the study.
Arm/Group | Diet Treatment | Standard Dose Saproterin Dihydrochloride | High Dose Saproterin Dihydrochloride
Number analyzed (Participants) | 7 | 7 | 7
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Diet Treatment | Standard Dose Saproterin Dihydrochloride | High Dose Saproterin Dihydrochloride
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT02677870/Prot_SAP_004.pdf
  • Informed Consent Form (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT02677870/ICF_003.pdf